CLINICAL TRIAL: NCT00041392
Title: PeriOperative Interventional Neuroprotection Trial (POINT)
Brief Title: Effects of Magnesium on Individuals Undergoing Coronary Artery Bypass Graft Surgery
Acronym: POINT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Pro00007128; R01HL069081 (NIH)
Record Dates: First submitted 2002-07-08; First posted 2002-07-09 (Estimated); Results first posted 2012-10-30 (Estimated); Last update posted 2013-07-30 (Estimated); Status verified 2012-04

CONDITIONS: Coronary Disease; Heart Diseases; Cardiovascular Diseases; Neurologic Manifestations
MeSH Terms: conditions — Coronary Disease; Heart Diseases; Cardiovascular Diseases; Neurologic Manifestations | interventions — Magnesium; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Magnesium (Active Comparator): 100 mg/kg magnesium
  Interventions: Drug: Magnesium
- 0.9 % saline (Placebo Comparator): 100 mg/kg 0.9 % saline
  Interventions: Drug: 0.9% saline

INTERVENTIONS:
Drug: Magnesium — 100 mg/kg
  Arms: Magnesium
Drug: 0.9% saline — Placebo
  Arms: 0.9 % saline

SUMMARY:
The purpose of this study is to examine the effects of supplemental magnesium on the neurocognitive function of individuals undergoing coronary artery bypass graft (CABG) surgery.

DETAILED DESCRIPTION:
BACKGROUND:

Approximately 400,000 individuals undergo heart operations each year and cognitive impairment occurs frequently following surgery. An increasing number of these individuals are elderly and are particularly susceptible to cognitive dysfunction following surgery. Cognitive impairment is most notable in the early stages following heart surgery, but it may persist in some individuals. While many people think cognitive impairment is subtle, transient, or subclinical, perioperative decline is associated with 5-year cognitive deterioration and reduced quality of life. Multiple strategies, both clinical and pharmacological, have been proposed to reduce the central nervous system dysfunction associated with heart surgery. However, most strategies have been unsuccessful, met with limited success, or are unrealistic from a cost or risk-benefit ratio for the majority of people. This study will examine the effectiveness of supplemental magnesium at preventing the cognitive decline associated with heart surgery.

DESIGN NARRATIVE:

This study will examine the effect of supplemental magnesium on the neurocognitive function of individuals undergoing CABG surgery. The two hypotheses to be tested include the following: 1) therapeutic levels of magnesium reduce post-operative neurocognitive dysfunction after heart surgery; and 2) therapeutic magnesium levels protect quality of life through reduced cognitive dysfunction after heart surgery. This double-blind study will enroll 400 individuals and randomly assign them to either the treatment group, which will receive 100 mg/kg of magnesium, or to the control group. Anesthesia management will be standardized to minimize any impact that anesthesia may have on neurologic or neuropsychologic outcome. Neurocognitive testing will be conducted prior to surgery, and 6 weeks and 1 year following surgery.

ELIGIBILITY:
Inclusion Criteria:

* Coronary heart disease

Exclusion Criteria:

* Early dementia
* History of psychiatric illness

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 389 (Actual)
Dates: Start 2001-12; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark F. Newman, MD, Study Chair — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Derived] Mathew JP, White WD, Schinderle DB, Podgoreanu MV, Berger M, Milano CA, Laskowitz DT, Stafford-Smith M, Blumenthal JA, Newman MF; Neurologic Outcome Research Group (NORG) of The Duke Heart Center. Intraoperative magnesium administration does not improve neurocognitive function after cardiac surgery. Stroke. 2013 Dec;44(12):3407-13. doi: 10.1161/STROKEAHA.113.002703. Epub 2013 Oct 8. PMID 24105697

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Hospital and preoperative clinic
Period: Overall Study
Arm/Group | Magnesium | 0.9 % Saline
Started | 198 | 191
Completed | 198 | 191
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Magnesium | 0.9 % Saline | Total
Number analyzed (Participants) | 198 | 191 | 389
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 78 | 74 | 152
  >=65 years | 120 | 117 | 237
Age Continuous [Mean (Standard Deviation); unit: years] | 68.6 (8.4) | 68.4 (8.0) | 68.5 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 54 | 66 | 120
  Male | 144 | 125 | 269
Region of Enrollment [Number; unit: participants]
  United States | 198 | 191 | 389

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function
Description: To characterize cognitive function over time, while minimizing potential redundancy in the cognitive measures, a factor analysis was performed on the cognitive test scores from baseline. We chose a four-factor solution, which represents 4 cognitive domains: verbal memory, abstraction and visuo-spatial orientation (executive function), visual memory and attention and concentration. To quantify overall cognitive function, a baseline cognitive index was first calculated as the mean of the 4 preoperative domain scores. The cognitive index score has a mean of zero and standard deviation of 0.5. Thus, any positive score is above the mean, any negative score is below the mean, and a score of 0.5 represents 1 SD above the mean. A continuous change score was then calculated by subtracting the baseline from the 6-week cognitive index. Negative scores indicate decline and positive scores indicate improvement.
Time Frame: Measured at baseline and 6 weeks
Measure: Mean (Standard Deviation); unit: Continuous cognitive change score
Arm/Group | Magnesium | 0.9 % Saline
Number analyzed (Participants) | 198 | 191
Continuous cognitive change score | 0.07 (0.28) | 0.12 (0.28)

ADVERSE EVENTS:
Arm/Group | Magnesium | 0.9 % Saline
Serious Adverse Events (participants affected / at risk) | 37/198 | 32/191
Other Adverse Events (participants affected / at risk) | 137/198 | 109/191
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnesium (N=198) | 0.9 % Saline (N=191)
Fever (Immune system disorders) | 1 (2) | 1 (2)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 1 (2)
Ventricular tachycardia (Cardiac disorders) | 3 (4) | 1 (4)
Pacemaker placement (Cardiac disorders) | 4 (6) | 2 (6)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (2) | 1 (2)
Congestive heart failure (Cardiac disorders) | 1 (2) | 1 (2)
Hypotension (Cardiac disorders) | 4 (4) | 0 (0)
Cardiac death (Cardiac disorders) | 2 (3) | 1 (3)
GI bleed (Gastrointestinal disorders) | 1 (2) | 1 (2)
Small bowel obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Bleeding (Blood and lymphatic system disorders) | 8 (10) | 2 (10)
Reexploration for bleeding (Surgical and medical procedures) | 3 (6) | 3 (6)
Sternal wound infection (Infections and infestations) | 1 (2) | 1 (2)
Stroke (Nervous system disorders) | 5 (11) | 6 (11)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (5) | 3 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 (10) | 8 (10)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 8 (14) | 6 (14)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 3 (6)
Renal insufficiency (Renal and urinary disorders) | 4 (5) | 1 (5)
Renal failure (Renal and urinary disorders) | 3 (5) | 2 (5)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Magnesium (N=198) | 0.9 % Saline (N=191)
Renal Insufficiency (Renal and urinary disorders) | 12 | 4
Postoperative bleeding (Blood and lymphatic system disorders) | 11 | 8
Hypotension (Cardiac disorders) | 11 | 10
Anemia (Cardiac disorders) | 16 | 7
Atrial fibrillation (Cardiac disorders) | 78 | 66
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 9 | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No